CLINICAL TRIAL: NCT01023256
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Preliminary Clinical Activity and Immunogenicity of Multiple Doses of MOR103 Administered Intravenously to Patients With Active Rheumatoid Arthritis
Brief Title: Safety and Preliminary Efficacy of MOR103 in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MSC-1001
Record Dates: First submitted 2009-11-19; First posted 2009-12-02 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; GM-CSF; MOR103
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Otilimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: MOR103, experimental (Experimental): Biological: MOR103 0.3 mg/kg or placebo
  Interventions: Drug: MOR103
- Group 2: MOR103, experimental (Experimental): Biological: MOR103 1.0 mg/kg or placebo
  Interventions: Drug: MOR103
- Group 3: MOR103, experimental (Experimental): Biological: MOR103 1.5 mg/kg or placebo
  Interventions: Drug: MOR103

INTERVENTIONS:
Drug: MOR103 — MOR103 0.3 mg/kg or placebo iv x 4 doses
  Arms: Group 1: MOR103, experimental
Drug: MOR103 — MOR103 1.0 mg/kg or placebo iv x 4 doses
  Arms: Group 2: MOR103, experimental
Drug: MOR103 — MOR103 1.5 mg/kg or placebo iv x 4 doses
  Arms: Group 3: MOR103, experimental

SUMMARY:
GM-CSF is considered to have a key role in the initiation and progression of arthritic inflammation. The purpose of this study is to evaluate the safety, preliminary efficacy, pharmacokinetics, and immunogenicity of multiple doses of MOR103, a human antibody to GM-CSF, in patients with active rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic systemic inflammatory disease that affects 0.5% to 1% of the adult population world wide. RA primarily affects the joints and is characterized by chronic inflammation of the synovial tissue, which eventually leads to the destruction of cartilage, bone and ligaments and can cause joint deformity.

Pro-inflammatory cytokines, such as tumor necrosis factor-alpha (TNFα), interleukin (IL)-1, IL-6 and granulocyte macrophage colony stimulating factor (GM-CSF), which lead to the activation and proliferation of immune cells, are found to be increased in the inflamed joint. Several preclinical findings support an anti-GM-CSF therapy for RA.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis (RA) per revised 1987 ACR criteria
* Active RA: ≥3 swollen and 3 tender joints with at least 1 swollen joint in the hand, excluding the PIP joint
* CRP > 5.0 mg/L (RF and anti-CCP seronegative); CRP >2 mg/l (RF and/or anti-CCP seropositive)
* DAS28 ≤ 5.1
* Stable regimen of concomitant RA therapy (NSAIDs, steroids, non- biological DMARDs).
* Negative PPD tuberculin skin test

Exclusion Criteria:

* Previous therapy with B or T cell depleting agents other than Rituximab (e.g. Campath). Prior treatment with Rituximab, TNF-inhibitors, other biologics (e.g. anti-IL-1 therapy) and systemic immunosuppressive agents is allowed with a washout period.
* Any history of ongoing, significant or recurring infections
* Any active inflammatory diseases other than RA
* Treatment with a systemic investigational drug within 6 months prior to screening
* Women of childbearing potential, unless receiving stable doses of methotrexate or leflunomide
* Significant cardiac or pulmonary disease (including methotrexate- associated lung toxicity)
* Hepatic or renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman P Korolkiewicz, MD, PhD, Study Director — MorphoSys AG
Locations (5):
- MorphoSys Investigative sites, MorphoSys Investigative Sites, Bulgaria
- MorphoSys Investigative sites, MorphoSys Investigative Sites, Germany
- MorphoSys Investigative sites, MorphoSys Investigative Sites, Netherlands
- MorphoSys Investigative sites, MorphoSys Investigative Sites, Poland
- MorphoSys Investigative sites, MorphoSys Investigatíve Sites, Ukraine

REFERENCES:
- [Result] Behrens F, Tak PP, Ostergaard M, Stoilov R, Wiland P, Huizinga TW, Berenfus VY, Vladeva S, Rech J, Rubbert-Roth A, Korkosz M, Rekalov D, Zupanets IA, Ejbjerg BJ, Geiseler J, Fresenius J, Korolkiewicz RP, Schottelius AJ, Burkhardt H. MOR103, a human monoclonal antibody to granulocyte-macrophage colony-stimulating factor, in the treatment of patients with moderate rheumatoid arthritis: results of a phase Ib/IIa randomised, double-blind, placebo-controlled, dose-escalation trial. Ann Rheum Dis. 2015 Jun;74(6):1058-64. doi: 10.1136/annrheumdis-2013-204816. Epub 2014 Feb 17. PMID 24534756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and screened between January 19, 2010 and February 9, 2012 at rheumatology centers in Europe (Bulgaria, Germany, the Netherlands, Poland and Ukraine).
Pre-assignment Details: Subject eligibility was determined at the screening visit (up to 35 days before treatment initiation) and confirmed at baseline before the first dose on day 1.
Groups:
- MOR103 0.3 mg/kg: MOR103 0.3 mg/kg IV once weekly for 4 weeks (total of 4 doses)
- MOR103 1.0 mg/kg: MOR103 1.0 mg/kg IV once weekly for 4 weeks (total of 4 doses)
- MOR103 1.5 mg/kg: MOR103 1.5 mg/kg IV once weekly for 4 weeks (total of 4 doses)
- Pooled Placebo: All patients who were randomized to the placebo arms in the 3 study cohorts. Placebo was administered IV once weekly for 4 weeks (total of 4 doses)
Period: Overall Study
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Placebo
Started | 25 | 22 | 24 | 27
Completed | 21 | 19 | 23 | 22
Not Completed | 4 | 3 | 1 | 5
Not completed — Protocol Violation | 2 | 3 | 0 | 0
Not completed — Randomized but not treated | 1 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All baseline participants were included in baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Placebo | Total
Number analyzed (Participants) | 24 | 22 | 23 | 27 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (8.3) | 49.0 (12.7) | 53.0 (9.9) | 53.8 (12.7) | 53.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 18 | 19 | 75
  Male | 3 | 5 | 5 | 8 | 21
Region of Enrollment [Number; unit: participants]
  Poland | 8 | 4 | 3 | 8 | 23
  Ukraine | 0 | 4 | 13 | 7 | 24
  Bulgaria | 12 | 7 | 4 | 6 | 29
  Netherlands | 0 | 0 | 1 | 2 | 3
  Germany | 4 | 7 | 2 | 4 | 17
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.3 (3.6) | 26.1 (4.6) | 25.7 (4.7) | 26.3 (3.5) | 26.1 (4.1)
Disease Activity Score based on 28 joints and erythrocyte sedimentation rate (DAS28-ESR) [Mean (Standard Deviation); unit: units on a scale] — The Disease Activity Score is a measure of overall disease activity and was calculated using 28 joints (DAS28) and the erythrocyte sedimentation rate (ESR) as the acute phase reactant (0 = no disease activity; 9.3 = maximal disease activity). In the MOR103 1.0 mg/kg group, one patient had missing data so the mean was calculated on 21 patients.
  units on a scale | 4.88 (0.54) | 4.78 (0.66) | 4.87 (0.38) | 4.88 (0.41) | 4.86 (0.50)
Rheumatoid factor (RF) status [Number; unit: participants] — Defined as RF levels >13.9 IU/mL. One patient in the MOR103 1.0 mg/kg group and one patient in the pooled placebo group had missing data.
  participants
    RF positive | 21 | 19 | 19 | 25 | 84
    RF negative | 3 | 2 | 4 | 1 | 10
    Missing | 0 | 1 | 0 | 1 | 2
Prior medication with non-biologic disease-modifying antirheumatic drugs (DMARDs) [Number; unit: participants] — Medication with non-biologic disease-modifying drugs in the 3 months prior to screening
  participants
    Treated with prior non-biologic DMARDs | 18 | 15 | 20 | 21 | 74
    Not treated with prior non-biologic DMARDs | 6 | 7 | 3 | 6 | 22
Prior medication with tumor necrosis factor (TNF) inhibitors [Number; unit: participants] — Medication with tumour necrosis factor inhibitors in the 3 months prior to screening
  participants
    Treated with prior TNF inhibitors | 1 | 0 | 0 | 2 | 3
    Not treated with prior TNF inhibitors | 23 | 22 | 23 | 25 | 93
Concomitant medication with non-biologic disease-modifying antirheumatic drugs (DMARDs) [Number; unit: participants] — Concomitant medication with non-biologic disease-modifying antirheumatic drugs at baseline
  participants
    Treated with concomitant non-biologic DMARDs | 22 | 17 | 21 | 26 | 86
    Not treated with concomitant non-biologic DMARDs | 2 | 5 | 2 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Patients With Treatment-emergent or Serious Adverse Events
Description: Data on treatment-emergent adverse events (MedDRA version 13.0) were collected at each visit (weeks 1, 2, 3, 4, 5, 6, 8, 10, 13, and 16). For a list of serious adverse events and adverse events occurring at a frequency of >5 % (>1 patient) in any treatment group, please see the adverse events listing.
Time Frame: From the first dose through the 16-week visit
Population: All patients who received treatment.
Measure: Number; unit: percentage of participants
Groups:
- Pooled Active: All patients receiving MOR103 at any dose
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Active | Pooled Placebo
Number analyzed (Participants) | 24 | 22 | 23 | 69 | 27
percentage of participants
  Percentage with treatment-emergent adverse events | 54.2 | 63.6 | 65.2 | 60.9 | 44.4
  Percentage with serious adverse events | 4.2 | 0.0 | 0.0 | 1.4 | 3.7

2. Secondary Outcome: Change From Baseline in Mean Disease Activity Score-28 Joints (DAS28) at 4 Weeks
Description: The primary exploratory efficacy outcome was change from baseline in Disease Activity Score calculated using 28 joints (DAS28) and the erythrocyte sedimentation rate (ESR) as the acute phase reactant (0 = no disease activity; 9.3 = maximal disease activity).
Time Frame: Change from baseline to week 4 (1 week after last MOR103 dose)
Population: All treated patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Placebo
Number analyzed (Participants) | 24 | 22 | 23 | 27
units on a scale | -0.2 (1.1) | -1.1 (0.9) | -0.6 (0.7) | 0.2 (0.8)
Statistical Analysis 1: Comparison: MOR103 0.3 mg/kg vs Pooled Placebo; Test type: Superiority or Other; p = 0.095, ANCOVA — P values were derived from pairwise comparisons between each MOR103 group and the pooled placebo group based on an analysis of covariance (ANCOVA) model. P values < 0.05 were considered significant; The ANCOVA model included fixed effect terms for dose and the covariate C-reactive protein level at baseline
Statistical Analysis 2: Comparison: MOR103 1.0 mg/kg vs Pooled Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; The ANCOVA model included fixed effect terms for dose and the covariate C-reactive protein level at baseline
Statistical Analysis 3: Comparison: MOR103 1.5 mg/kg vs Pooled Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 2, analysis 1]; The ANCOVA model included fixed effect terms for dose and the covariate C-reactive protein level at baseline

3. Other Pre Specified Outcome: Change From Screening in Outcome Measures in Rheumatology (OMERACT)-Rheumatoid Arthritis Magnetic Resonance Imaging Studies Mean Sum Score for Synovitis at Week 4
Description: Magnetic resonance imaging (MRI) was performed on the wrist and hand on the side with the most swollen joints (or the right side if swollen joints were equivalent). The 2nd to 5th metacarpophalangeal joints and 3 wrist joints (distal radioulnar, radiocarpal, and intercarpal-carpometacarpal joints) were scored on a scale of 0 = no synovitis to 3 = severe synovitis. MRIs were scored by 2 independent experts blinded to patient data and chronology. The sum score is the average of the 2 reader scores for each of the 7 joints. The range of the sum score is thus 0 = no synovitis in any joint to 21 = severe synovitis in all joints.
Time Frame: Change from screening to week 4 (1 week after last MOR103 dose)
Population: At week 4, MRI data were not available for 5 placebo patients, 2 MOR103 0.3 mg/kg patients, 2 MOR103 1.0 mg/kg patients, and 1 MOR103 1.5 mg/kg patient.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Placebo
Number analyzed (Participants) | 22 | 20 | 22 | 22
units on a scale | -0.37 (3.09) | -1.50 (2.87) | -0.50 (2.22) | -0.66 (3.09)

4. Secondary Outcome: Change From Baseline in Mean Disease Activity Score-28 Joints (DAS28) at 8 Weeks
Description: as for outcome 2
Time Frame: Change from baseline to week 8 (5 weeks after last MOR103 dose)
Population: All treated patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Placebo
Number analyzed (Participants) | 24 | 22 | 23 | 27
units on a scale | -0.3 (0.9) | -1.0 (1.3) | -0.6 (0.9) | -0.1 (0.9)
Statistical Analysis 1: Comparison: MOR103 0.3 mg/kg vs Pooled Placebo; Test type: Superiority or Other; p = 0.421, ANCOVA — [p-value comment as in outcome 2, analysis 1]; The ANCOVA model included fixed effect terms for dose and the covariate C-reactive protein level at baseline
Statistical Analysis 2: Comparison: MOR103 1.0 mg/kg vs Pooled Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 2, analysis 1]; The ANCOVA model included fixed effect terms for dose and the covariate C-reactive protein level at baseline
Statistical Analysis 3: Comparison: MOR103 1.5 mg/kg vs Pooled Placebo; Test type: Superiority or Other; p = 0.065, ANCOVA — [p-value comment as in outcome 2, analysis 1]; The ANCOVA model included fixed effect terms for dose and the covariate C-reactive protein level at baseline

5. Secondary Outcome: Percentages of Subjects With American College of Rheumatology 20% Improvement (ACR20) at Week 4
Description: The percentage of patients achieving an ACR20 response (20% improvement based on ACR improvement criteria) in each group. ACR20 improvement criteria require at least 20% improvement in both swollen and tender joints counts and 3 out of 5 of the following parameters: pain visual analog scale, patient global assessment, physician global assessment, acute phase reactant (erythrocyte sedimentation rate or C-reactive protein), and functional questionnaire.
Time Frame: Week 4 (1 week after last MOR103 dose)
Population: All participants were included in ACR response calculations. Patients lacking data required for calculation of an ACR response were considered as not having an ACR response. 1 patient in the MOR103 0.3 mg/kg group, 1 patient in the MOR103 1.0 mg/kg group, and 5 patients in the pooled placebo group had missing data for ACR calculations.
Measure: Number; unit: percentage of participants
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Placebo
Number analyzed (Participants) | 24 | 22 | 23 | 27
percentage of participants | 25.0 | 68.2 | 30.4 | 7.4
Statistical Analysis 1: Comparison: MOR103 0.3 mg/kg vs Pooled Placebo; Test type: Superiority or Other; p = 0.243, Fisher Exact — P values <0.05 were considered to be statistically significant; Patients with missing values were not included
Statistical Analysis 2: Comparison: MOR103 1.0 mg/kg vs Pooled Placebo; Test type: Superiority or Other; p < 0.0001, Fisher Exact — P values < 0.05 were considered significant; Patients with missing values were not included
Statistical Analysis 3: Comparison: MOR103 1.5 mg/kg vs Pooled Placebo; Test type: Superiority or Other; p = 0.135, Fisher Exact — P values <0.05 were considered to be statistically significant; Patients with missing values were not included

6. Secondary Outcome: Change From Baseline in Mean Swollen and Tender Joint Counts at Weeks 4 and 8
Description: Swollen joint counts were based on 66 joints and tender joint counts were based on 69 joints.
Time Frame: Change from baseline to week 4 (1 week after last MOR103 dose) and change from baseline to week 8
Population: All treated patients
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Placebo
Number analyzed (Participants) | 24 | 22 | 23 | 27
joints
  Change in swollen joint count at week 4 | -1.7 (2.4) | -3.5 (5.1) | -3.3 (3.2) | 0.1 (3.5)
  Change in swollen joint count at week 8 | -1.9 (2.2) | -4.1 (4.4) | -3.3 (3.1) | -0.8 (3.6)
  Change in tender joint count at week 4 | 0.1 (7.1) | -4.8 (3.2) | -3.7 (6.2) | 2.0 (6.4)
  Change in tender joint count at week 8 | 0.3 (5.0) | -6.8 (4.1) | -4.0 (5.3) | 2.1 (8.0)

7. Secondary Outcome: Change From Baseline in Patient-reported Outcomes at Weeks 4 and 8
Description: Patient-reported outcomes included patient's self-assessment of pain (measured on a 100 mm visual analogue scale [VAS] from 0 = best to 100 = worst), the Health Assessment Questionnaire-Disability Index (HAQ-DI; 0 = best to 3 = worst), the patient's global assessment of disease activity (measured on a 100 mm visual analogue scale [VAS] from 0 = best to 100 = worst), and fatigue, which was measured by the Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue self-assessment scale (0 = worst; 52 = best).
Time Frame: Change from baseline at week 4 (1 week after last MOR103 dose) and change from baseline at week 8
Population: All treated patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Placebo
Number analyzed (Participants) | 24 | 22 | 23 | 27
units on a scale
  Change in pain at week 4 | -8.6 (22.8) | -17.4 (17.2) | -11.4 (11.5) | -3.3 (16.5)
  Change in pain at week 8 | -4.1 (23.1) | -13.4 (20.9) | -9.5 (11.9) | -8.0 (16.1)
  Change in HAQ-DI at week 4 | -0.21 (0.41) | -0.53 (0.52) | -0.31 (0.24) | -0.45 (0.54)
  Change in HAQ-DI at week 8 | -0.21 (0.56) | -0.51 (0.56) | -0.25 (0.22) | -0.44 (0.54)
  Change in patient global assessment at week 4 | -2.7 (20.5) | -16.6 (15.6) | -6.0 (17.7) | -3.0 (16.1)
  Change in patient global assessment at week 8 | -4.5 (21.9) | -13.3 (24.7) | -4.0 (8.3) | -8.2 (17.5)
  Change in FACIT fatigue score at week 4 | 2.7 (9.2) | 9.1 (10.2) | 3.1 (6.0) | 3.0 (8.1)
  Change in FACIT fatigue score at week 8 | 2.1 (5.6) | 9.4 (12.6) | 4.7 (7.1) | 4.3 (9.1)

8. Other Pre Specified Outcome: Change From Screening in Outcome Measures in Rheumatology (OMERACT)-Rheumatoid Arthritis Magnetic Resonance Imaging Studies Mean Sum Score for Synovitis at Week 8
Description: as for outcome 3
Time Frame: Change from screening to week 8
Population: At week 8, MRI data were not available for 6 placebo patients, 5 MOR103 0.3 mg/kg patients, 1 MOR103 1.0 mg/kg patient, and 2 MOR103 1.5 mg/kg patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Placebo
Number analyzed (Participants) | 19 | 21 | 21 | 21
units on a scale | -0.48 (3.49) | -0.90 (2.83) | -1.00 (2.73) | -0.91 (3.06)

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events reported from the time of the first dose of MOR103 or placebo to the end of the 16-week follow up period.
Groups:
- Pooled Placebo: Pooled placebo group included all patients who were randomized to placebo in the 3 study cohorts. Placebo was administered IV once weekly for 4 weeks (total of 4 doses)
Arm/Group | MOR103 0.3 mg/kg | MOR103 1.0 mg/kg | MOR103 1.5 mg/kg | Pooled Active | Pooled Placebo
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/22 | 0/23 | 1/69 | 1/27
Other Adverse Events (participants affected / at risk) | 11/24 | 22/22 | 14/23 | 47/69 | 12/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOR103 0.3 mg/kg (N=24) | MOR103 1.0 mg/kg (N=22) | MOR103 1.5 mg/kg (N=23) | Pooled Active (N=69) | Pooled Placebo (N=27)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOR103 0.3 mg/kg (N=24) | MOR103 1.0 mg/kg (N=22) | MOR103 1.5 mg/kg (N=23) | Pooled Active (N=69) | Pooled Placebo (N=27)
Nasopharyngitis (Infections and infestations) | 1 (2) | 7 (7) | 1 (1) | 9 (10) | 3 (3)
Viral respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 2 (3) | 9 (10) | 0 (0) — Worsening or flares of rheumatoid arthritis. In 8 of the 9 MOR103 subjects with RA exacerbations, this AE occurred after the last dose of MOR103 (10 days to >12 weeks), suggesting that disease flares were related to withdrawal of active treatment.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (5) | 1 (1) | 6 (7) | 1 (1)
Edema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Carbon monoxide diffusing capacity decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — Based on investigator reports of clinically relevant events.
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) — Includes patients with preferred term "rash" and preferred term "rash maculo-papular"
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Key limitations of this trial include its small sample size, limited duration, and exclusion of patients with severe rheumatoid arthritis. Larger clinical trials are needed to confirm these data and define the optimal MOR103 dosage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information supplied by MorphoSys is considered confidential until publication and shall not be disclosed without prior written consent from MorphoSys. No data can be published in any format without prior approval of the MSC-1001 Publication Committee, which has final decision on approving submissions for publication. In the event of disagreement in the content of a publication, both the Author's and MorphoSys' opinion will be fairly and sufficiently represented in the publication.